CLINICAL TRIAL: NCT00225095
Title: A Phase I/II, Randomized, Controlled, Double Blind, Study of Chondrogen - Adult Universal Cell Delivered by Intra-Articular Injection Following Meniscectomy in Patients 18-60 Years
Brief Title: A Phase I/II Study of Chondrogen Delivered by Intra-Articular Injection Following Meniscectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mesoblast International Sàrl (Industry)
Collaborators: University of Southern California (Other); Midwest Orthopedics at Rush - Chicago, IL (Unknown); Unlimited Research - San Antonio, TX (Unknown); Triangle Orthopaedic Associates, P.A. (Other); Orthopedic Center of Vero Beach - Vero Beach, FL (Unknown); OrthoIndy (Other); TRIA Orthopaedic Center (Other); Greater Chesapeake Orthopaedic Associates, LLC (Other)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Osiris 550
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Recovery Following Partial Medial Meniscectomy
Keywords: meniscectomy; Chondrogen; Mesenchymal Stem Cells; Osiris
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Chondrogen - dose 1 (Active Comparator): Chondrogen - 50 million cells
  Interventions: Drug: Mesenchymal Stem Cells
- Chondrogen - dose 2 (Active Comparator): Chondrogen - 150 million cells
  Interventions: Drug: Mesenchymal Stem Cells
- Vehicle Control (Other): Vehicle Control
  Interventions: Drug: Hyaluronan

INTERVENTIONS:
Drug: Mesenchymal Stem Cells
  Arms: Chondrogen - dose 1; Chondrogen - dose 2
Drug: Hyaluronan
  Arms: Vehicle Control

SUMMARY:
The purpose of this study is to determine whether Chondrogen is a safe and effective post-operative treatment of the knee following menisectomy (the surgical removal of all or part of a torn meniscus).

DETAILED DESCRIPTION:
Chondrogen is a preparation of adult mesenchymal stem cells (MSCs) in a solution containing hyaluronic acid. Preclinical studies have shown that injection of Chondrogen aids in the repair of meniscal tissue following meniscectomy. In Chondrogen treated subjects, surgically removed meniscal tissue was regenerated, cartilage surface was protected, and joint damage was decreased in comparison to control subjects. These benefits persisted at least one year.

Three groups of recent meniscectomy patients will be followed in this study, including patients that will receive placebo and patients that will be treated with one of two possible doses of Chondrogen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60, inclusive
* In need of medial meniscectomy
* Normal axial alignment
* Stable knee- previous ligament reconstruction, if stable
* Removal of at least 50% of the affected portion of the medial meniscus
* Intact articular cartilage in posterior meniscal weight-bearing zone
* Willingness to follow normal post-operative rehabilitation
* Willingness to participate in follow-up for two years from the time of meniscectomy surgery
* Ability to understand and willingness to sign consent form

Exclusion Criteria:

* Pregnant or lactating
* ACL or other support structure damage confirmed at surgery
* Grade III or IV cartilage damage (Cartilage loss greater than 50% thickness in area >15mm on weight-bearing aspect of femoral condyle or tibial plateau)
* Synvisc, steroid, or corticosteroid injections in preceding 3 months
* Diffuse synovitis at time of arthroscopy
* Inflammatory arthritis
* Oral steroid, methotrexate therapy
* Unable to follow post-operative exercise regimen or return for evaluations
* Active alcohol or substance abuse within 6 months of study entry
* Current and active tobacco product use
* Patient is positive for HIV
* Patient is positive for hepatitis (past history of Hepatitis A is allowed)
* Any medical condition, which in the opinion of the clinical investigator, would interfere with the treatment or outcome of the patient
* Indwelling pacemaker
* Cerebral aneurysm clips
* Ear, eye and penile implants with avian components
* Electrical indwelling device such as bone stimulator
* Indwelling magnets as tissue expander for future implants
* Known allergy to avian, bovine or porcine protein

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Meniscal Volume | 6 months
  Changes in meniscal volume over the course of the study as determined by MRI

SECONDARY OUTCOMES:
Quality of Life Questionnaire | 2 years
  Determination of Quality of Life will be measured by the KOOS instrument (Knee injury and Osteoarthritis Outcome Score).
Visual Analog Scale (VAS) | Baseline to 2 years
  Patient perception of pain will be documented using a single VAS pain scale.
Lysholm Knee Scale | 2 years
  Lysholm knee score will be determined according to the questionnaire
Safety Assessment Adverse Event | 2 years
  Number of participants with Adverse Events.
Safety Assessment Immunological | 2 years
  Number of participants with clinically significant abnormalities in immunological measures
Safety Assessment Laboratory | 2 years
  Number of participants with clinically significant abnormalities in laboratory assessments
Safety Assessment Physical Exam | 2 years
  Number of participants with clinically significant abnormalities in physical examinations.
Safety Assessment Magnetic Resonance Imaging (MRI) | 2 years
  Number of participants with clinically significant abnormalities in Magnetic Resonance Imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Williams, Ph.D., Study Director — Osiris Therapeutics, Inc.
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - Orthopedic Center of Vero Beach, Vero Beach, Florida
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - Ortholndy, Indianapolis, Indiana
  - Greater Chesapeake Associates, Baltimore, Maryland
  - TRIA Orthopaedic Center, Bloomington, Minnesota
  - Triangle Orthopaedics Associates, P.A., Durham, North Carolina
  - Unlimited Research, San Antonio, Texas

REFERENCES:
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Murphy JM, Fink DJ, Hunziker EB, Barry FP. Stem cell therapy in a caprine model of osteoarthritis. Arthritis Rheum. 2003 Dec;48(12):3464-74. doi: 10.1002/art.11365. PMID 14673997
- [Derived] Vangsness CT Jr, Farr J 2nd, Boyd J, Dellaero DT, Mills CR, LeRoux-Williams M. Adult human mesenchymal stem cells delivered via intra-articular injection to the knee following partial medial meniscectomy: a randomized, double-blind, controlled study. J Bone Joint Surg Am. 2014 Jan 15;96(2):90-8. doi: 10.2106/JBJS.M.00058. PMID 24430407
- See also: Osiris Therapeutics, Inc. Home Page — http://www.osiristx.com